CLINICAL TRIAL: NCT06129994
Title: Ecological Momentary Assessment Study of Adolescents and Young Adults With Type 1 Diabetes (EMA-T1D)
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Jennifer Iyengar, Clinical Assistant Professor, University of Michigan
Other Study IDs: HUM00234964
Record Dates: First submitted 2023-10-30; First posted 2023-11-13 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Optional serum and plasma biospecimens retained for the purpose of future research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Group: Participants will complete the observational study over the 15 day study period
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Participants will complete an in-person baseline study visit with fasting blood draw, medical and health history, anthropometrics and vital signs, and surveys. If participants are not currently using a CGM, one will be placed. The LifeData study mobile app will be installed on the participant's smartphone. Over the two-week home monitoring period, participants will be asked to wear the CGM and respond to EMA questions three times daily. After the end of the home monitoring period, a remote visit will be performed in which the CGM will be removed by the study participant at home; the study team will obtain all data available from the CGM and insulin pump (if available); and surveys will be collected.

SUMMARY:
This single site investigator-initiated prospective observational study will enroll up to 150 participants 13-26 years of age with Type 1 diabetes (T1D) and utilize ecological momentary assessment methods (EMA) to examine associations between different diabetes psychological domains (distress, anxiety, and depression) in real-time on self-efficacy, self-management behaviors, and glycemic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes for at least six months
* Fluent in spoken and written English
* Willing to carry around their mobile phone during the home monitoring period with daily access to cellular or WiFi connectivity
* Willing to wear a continuous glucose monitor (CGM) device during the home monitoring period

Exclusion Criteria:

* Any social or medical condition that would, in the opinion of the Principal Investigator (PI), prevent complete participation in the study or would pose significant hazard to the subject's participation
* Skin conditions or diseases that would interfere with the CGM sensor placement or accuracy (such as extensive psoriasis, extensive eczema, scarring, etc.)
* Scheduled X-ray, MRI, CT scan, or high-frequency electrical heat (diathermy) treatment during the period of CGM wear (or any other activity that would necessitate CGM sensor or insulin pump removal) that cannot be scheduled around or accommodated within the study assessment windows
* Currently pregnant or plan to become pregnant during participation in the study

Ages: 13 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants must meet eligibility criteria to be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-08-10 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
Ecological Momentary Assessment (EMA) methods for measuring diabetes distress | Home monitoring (days 1-14)
  Diabetes distress score via EMA
Ecological Momentary Assessment (EMA) methods for measuring anxiety | Home monitoring (days 1-14)
  Anxiety score via EMA
Ecological Momentary Assessment (EMA) methods for measuring depression | Home monitoring (days 1-14)
  Depression score via EMA

SECONDARY OUTCOMES:
Glycemic Outcomes | Home monitoring (days 1-14)
  Percent Time in range (70-180mg/dl), Percent time with low glucose readings (<70mg/dl), Percent time with high glucose (>180mg/dl)
Hemoglobin A1c | Baseline
  Hemoglobin A1c

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Iyengar, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No